CLINICAL TRIAL: NCT04510727
Title: Using OCT Imaging to Determine the Presence of Residual Tumor Cells After C&D for Superficial and Nodular BCC: A Prospective Study.
Brief Title: Optical Coherence Tomography Guided C&D
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: device not available to initiate study.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Keyvan Nouri, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20200212
Record Dates: First submitted 2020-08-09; First posted 2020-08-12 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Basal Cell Carcinoma
Keywords: Superficial basal cell carcinoma; Nodular basal cell carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Tomography, Optical Coherence; Curettage; Desiccation; Dilatation and Curettage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- OCT Guided C&D Group (Experimental): Participants in this group will receive OCT imaging immediately prior, immediately after and 2 months after post standard of care C&D.
  Interventions: Device: Optical Coherence Tomography (OCT); Procedure: Curettage & Desiccation (C&D) Procedure

INTERVENTIONS:
Device: Optical Coherence Tomography (OCT) — VivoSight Dx OCT system from Michelson Diagnostics Ltd. OCT will be used to visualize the tumor and lesion in the skin.
Procedure: Curettage & Desiccation (C&D) Procedure — Standard of care C&D where the basal cell carcinoma lesion will be scraped to its base using a Fox dermal curette and an electrodesiccation machine.

SUMMARY:
The purpose of the study is to identify the presence of residual superficial and nodular basal cell carcinoma (BCC) status-post curettage and desiccation (C&D) by using optical coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

* Patients of any: age, gender, Fitzpatrick skin type and ethnicity.
* Primary BCC of any type, except aggressive types that fit the criteria for Mohs surgery
* No prior treatment on the lesion within the last 3 months.
* Lesions anywhere except the head, neck and distal extremities.
* Willing and able to sign informed consent

Exclusion Criteria:

* Aggressive BCC types.
* Recurrent tumors.
* Lesion treated within last 3 months.
* Lesions on head and neck (high risk areas)
* Lesions on distal extremities (thin epidermis not preferred for OCT).
* Pregnant women.
* Patients less than 18 years old.
* Prisoners.
* Any other condition or circumstance that, in the opinion of the Investigator, may compromise the subject's ability to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of residual basal cell carcinoma tumor cells | 2 months (post C&D procedure)
  The incidence of residual superficial and nodular basal cell carcinoma tumor cells after standard of care C&D as assessed using the OCT.

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Nouri, MD, Principal Investigator — University of Miami
Locations (1):
- Maria V Muniz, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No